CLINICAL TRIAL: NCT04836936
Title: Auriculotherapy in the Treatment of Pre-Operative Anxiety - A Randomized, Prospective, Placebo-Controlled Clinical Trial
Brief Title: Auriculotherapy in the Treatment of Pre-Operative Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor of Anesthesiology (with Tenure) and Orthopedic Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20120027
Record Dates: First submitted 2021-03-09; First posted 2021-04-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Preoperative
Keywords: Nephrectomy; Auriculotherapy

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-Controlled trial involving patients undergoing partial or total nephrectomy.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The only person unblinded to treatment allocation will be the Principal investigator or individual who will perform the auriculotherapy treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Auriculotherapy cryopuncture device without nitrogen gas (Placebo Comparator): Auriculotherapy will be performed in the pre-operative setting by PI or trained designee using an empty cryopuncture device without nitrogen gas. The patient will otherwise receive standard of care treatment for surgery and post-operative pain management.
  Interventions: Device: Auriculotherapy cryopuncture device without nitrogen gas
- Auriculotherapy cryopuncture device with nitrogen gas (Active Comparator): Auriculotherapy will be performed in the pre-operative setting by PI or trained designee using a cryopuncture device with nitrogen gas. The patient will otherwise receive standard of care treatment for surgery and post-operative pain management.
  Interventions: Device: Auriculotherapy cryopuncture device with nitrogen gas

INTERVENTIONS:
Device: Auriculotherapy cryopuncture device without nitrogen gas — Auriculotherapy cryopuncture device without nitrogen gas will be administered. Application of this placebo device will be performed in the same manner as the treatment, but without the expulsion of nitrogen gas.
  Arms: Auriculotherapy cryopuncture device without nitrogen gas
Device: Auriculotherapy cryopuncture device with nitrogen gas — Auriculotherapy cryopuncture device with nitrogen gas will be administered. The tip of the cryopuncture will be sanitized and placed on each treatment point of the ear, releasing a spurt of nitrogen gas for 2 seconds on each point (6 points total).
  Arms: Auriculotherapy cryopuncture device with nitrogen gas

SUMMARY:
The goal of this clinical trial is to use the validated PROMIS Emotional Distress - Anxiety - Short Form 8a and PROMIS Emotional Distress-Depression-Short Form pre-and post-intervention to establish a superior correlation between the auriculotherapy treatment and the reduction of perioperative anxiety. Subject population will include those having a partial or total nephrectomy for cancer. Drawing the role that auriculotherapy may play in reducing perioperative anxiety related requirement after surgery may also help in reducing the risk of opioid use disorders (OUD) since anxiety has been found to be a major risk factor for OUD in surgical patients. Therefore, this trial will also examine the effect of the auriculotherapy intervention in reducing opioid requirement after surgery.

DETAILED DESCRIPTION:
Sixty subjects undergoing total or partial nephrectomies will be asked to participate in this IRB approved placebo-controlled randomized study. Potential subjects will be recruited out of the surgeon's office or at a preoperative clinical visit prior to surgery. The clinical care team will introduce the study and request permission for the research team to speak with the patient. If the subject agrees to be approached by a member of the research team, then the research team will approach the subject. During the Informed Consent, a PI or Co-I will be available to answer final questions and facilitate the process.

After signing an informed consent, the subjects will be equally randomized to either active auriculotherapy treatment (with nitrogen gas) or placebo auriculotherapy treatment (without nitrogen gas). Each subject will be asked to complete the PROMIS Emotional Distress - Anxiety - Short Form 8a, the PROMIS Emotional Distress-Depression-Short Form and Pain Catastrophizing Scale (PCS) in the pre-operative setting. Those whose anxiety scores are ≥19 and ≤29 will be included in the study and randomly distributed to either treatment allocation.

Randomization will occur by assigning the participant a subject ID number, and this ID number will correspond to a treatment allocation based on a pre-designed randomization schema. This treatment allocation (intervention/control) will be contained in a sealed, opaque, envelope with the subject ID number that is designated on envelope. The master randomization list will be created and held by an independent data monitor who will both create and hold the master randomization list. A data manager research associate will confidentially reveal the randomization to the PI or Amy Monroe so that the study coordinators, Co-Is and subjects will be blinded. PI or Amy Monroe, and the data managing associate will be the only individuals who are unblinded.

Study assessments will be conducted on the day of surgery, in the pre-operative setting. This will include the PROMIS Emotional Distress - Anxiety - Short Form 8a as this is the first assessment conducted after obtaining Informed Consent. It is used to assess eligibility for the study. This assessment will take roughly 5 minutes.

Auriculotherapy treatment will also occur in the pre-operative setting, within one hour of surgery and after the patient has received a peripheral nerve block. For the active treatment group, a nitrogen gas canister will be applied to a cryopuncture device (manual attached), and the tip of the cryopuncture will be sanitized and placed on each treatment point of the ear, releasing a spurt of gas for 2 seconds on each point (7 points total). For the sham device, an empty canister will be applied to the cryopuncture device, and in exactly the same fashion as the treatment group, the tip of the cryopuncture will be sanitized and placed on each treatment point of the ear. Instead of releasing a spurt of nitrogen gas, the empty canister will make the same noise as a full canister, but without the expulsion of gas. We are not expecting any adverse events from performing this technique. The only "adverse event" that is expected is a mild local blistering/scab, which may occur within 24 hours after the treatment. In our experience in our ongoing auriculotherapy study (24 subjects enrolled), we did not observe this adverse event. In the experience of Dr. Chelly(11 years) and Dr. Alimi (30 years), any local blistering or ulceration is extremely mild, and resolves in days without any intervention. No potential adverse effect would require immediate treatment or delay the surgery.

After surgery, the subject will be assessed for pain medication requirement and pain scores in the post-anesthesia care unit (PACU) and then assessed daily until discharge. Upon discharge, subjects will repeat the PROMIS Emotional Distress questionnaires and the PCS. Additionally, subjects will be asked to complete an overall satisfaction questionnaire measured on a scale to 0-10.

The subjects will take home a diary where they will record daily NRS pain scores (scale 0-10), daily anxiety level (scale 0-10) and daily analgesic/opioid requirement for one-week post-op. The subject will be contacted daily after discharge until completion of the pain diary at Day 7 post-op, and will also be contacted once at 30-day and 90-day post-op to report the PROMIS Emotional Distress -Anxiety- Short Form 8a, the PROMIS Emotional Distress-Depression-Short Form, and Pain Catastrophizing Scale (PCS) verbally over the telephone. The subject will be contacted via phone daily to gather their responses post op to the surveys, a maximum of three times. If we are unable to reach the subject after 3 days they will be considered lost to follow up. If In addition to this, the subject will be asked to assess their functional recovery using the SF-12 questionnaire, and to report their VAS pain score/opioid consumption for the previous week.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Scheduled to undergo partial or full elective nephrectomy
* Subject is willing and able to provide informed consent
* Anxiety score ≥ 19 and ≤ 29 on the PROMIS Emotional Distress-Anxiety-Short Form 8a.

Exclusion Criteria:

* Opioid dependence, based on the DSM definition of Opioid Use Disorder (OUD)
* Chronic pain condition where daily opioid use is needed
* History of fibromyalgia
* Anatomical malformation of ear (genetic or trauma-induced)
* Vasculopathy of ear
* Raynaud's disease
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Day of surgery through discharge or post-operative day 30, whichever came first
  Demonstrate how auriculotherapy using the cryopuncture device changes participant's total opioid consumption following nephrectomy surgery.

SECONDARY OUTCOMES:
Pre-operative emotional distress related to anxiety | Screening visit
  Pre-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire prior to surgery. There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative emotional distress related to anxiety | Day of surgery through 3 months post-operative
  Post-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire.There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Pre-operative emotional distress related to depression | Screening visit
  Pre-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire prior to surgery. There are 8 questions about how the participant many have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative emotional distress related to depression | Day of surgery through 3 months post-operative
  Post-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire. There are 8 questions about how the participant many have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Pre-operative pain rating using the Pain Catastrophizing Scale | Screening visit
  Pre-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome.
Post-operative pain rating using the Visual Analog Scale (VAS) | Day of surgery through 3 months post-operative
  Post-operative pain ratings will be measured by the assessment of the participant's answers to the Visual Analog Scale (VAS). This measurement is a visual scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. The participant will be asked to score pain at its best and worst over the period since they were last asked. Higher scores present a worse outcome.
Post-operative pain rating using the Pain Catastrophizing Scale | Day of surgery through 3 months post-operative
  Post-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome.
Post-operative analgesic utilization | Day of surgery through 3 months post-operative
  Post-operative analgesic utilization will be measured using electronic medical records and patient-recorded diaries of daily analgesic/opioid requirements.
Functional Recovery | Day of surgery through 3 months post-operative
  Functional recovery will be measured by the assessment of the participant's answers to the Functional Recovery Questionnaire 12-Item Short Form Health Survey (SF-12). The SF-12 Health Survey includes questions from the SF-36 Health Survey (Version 1).These include: 2 questions concerning physical functioning; 2 questions on role limitations because of physical health problems; 1 question on bodily pain; 1 question on general health perceptions; 1 question on vitality (energy/fatigue); 1 question on social functioning; 2 questions on role limitations because of emotional problems; and 2 questions on general mental health (psychological distress and well-being). Overall score can range from 12 to 53. Higher scores present a better outcome.
Overall patient satisfaction | Day of surgery through discharge or post-operative day 30, whichever came first
  Participants will be asked to assess their overall satisfaction upon discharge on a scale of 0 (least satisfaction) to 10 (highest satisfaction) at the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No